CLINICAL TRIAL: NCT04048018
Title: Performance Evaluation of the VIDAS TB-IGRA Assay.
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: B2694-CTPR
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Active Tuberculosis; Latent Tuberculosis Infection; Non-Tuberculous Mycobacterial (NTM) Pneumonia
Keywords: Interferon Gamma Release Assay; Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis; Pneumonia; Tuberculosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Active Tuberculosis Patient
  Interventions: Diagnostic Test: Blood draw and IGRA test
- High risk for LTBI Participant
  Interventions: Diagnostic Test: Blood draw and IGRA test
- Low risk for prior TB infection Participant
  Interventions: Diagnostic Test: Blood draw and IGRA test
- NTM patient
  Interventions: Diagnostic Test: Blood draw and IGRA test
- Precision patient
  Interventions: Diagnostic Test: Blood draw and IGRA test

INTERVENTIONS:
Diagnostic Test: Blood draw and IGRA test — One to two blood samples will be obtained from participants in all arms in order to conduct testing.

SUMMARY:
This study will evaluate the performance of the VIDAS® Interferon Gamma (IFN-γ) Release Assay (TB-IGRA) assay, which is intended for use as an aid in the diagnosis of tuberculosis infection. This study is designed to assess (1) the sensitivity of this assay, (2) its percent agreement with other diagnostic tests, (3) its measurement precision , and (4) any potential interference of the presence of other non-tuberculosis mycobacterial bacterial infections with this assay.

DETAILED DESCRIPTION:
Tuberculosis (TB) infection is one of the top 10 causes of death in the world and the leading cause of death due to a single infectious agent. Millions of people are infected with TB each year which can pose significant economic and health care burdens on the global population.

TB can infected the lungs (pulmonary TB) or other organs such as the brain, and kidneys (extra-pulmonary TB). When a person with pulmonary TB coughs or sneezes, water droplets containing M. tuberculosis are expelled into the air. Persons can become infected with TB when they inhale air containing these water droplets, however, not everyone infected with Mycobacterium tuberculosis (Mtb) becomes ill. Therefore two TB-related conditions exist: latent TB infection (LTBI) and TB disease.

People with latent TB infection are not ill and do not present TB symptoms or have TB disease. The only sign of TB infection is a positive reaction to the tuberculin skin test or TB blood tests such as IGRA tests. People with latent TB infection are not contagious and cannot spread TB infection to others.

Identification and treatment of LTBI can substantially reduce the risk of developing active disease. However, there is no diagnostic gold standard for LTBI. Two types of test are currently available for the identification of LTBI: the tuberculin skin test (TST) and the TB Interferon Gamma (IFN-γ) Release Assay (TB-IGRA). Evidence suggests that both TST and TB-IGRA are acceptable but not perfect because they detect indirect markers of Mtb exposure and indicate a cellular immune response to M. tuberculosis. TB-IGRAs have a number of advantages compared to TST which promote their progressive adoption in the clinical practice and in guidelines.

ELIGIBILITY:
Active TB Population

Inclusion Criteria:

A person classified as or suspected of having M. tuberculosis disease (active TB):

A person with known HIV status, determined by a laboratory or rapid test performed no earlier than one month prior to, or at the time of inclusion into this study A person of age ≥ 2 years

Exclusion Criteria:

A person who has been on an anti-TB treatment for >15 days for the ongoing infection Pregnant women A person who has received an anti-tumor necrosis factor (TNF) alpha treatment within the previous 3 months A person who has had prior TST A person with an NTM infection A person with positive HIV status.

High Risk for TB infection

Inclusion criteria :

A person who is at increased risk for M. tuberculosis infection (and therefore LTBI) and/or for progression to active TB:

A person with age ≥ 2 years A person with known HIV status

Non-inclusion criteria will be:

A person who has or has had active TB A person who has received treatment for active TB or LTBI A person who has received an anti-TNF alpha treatment A person who has had a TST Pregnant women Person who has been an NTM infection

Low Risk for TB Infection

Inclusion criteria

Generally healthy people, unlikely to have encountered TB disease in the past, that may be subject to TB testing for professional, academic or personal reasons (e.g.: students, healthcare personnel and healthcare volunteers, military recruits) A person with age ≥ 18 years old

Non-inclusion criteria A person who is considered at high risk for LTBI A person who has or has had active TB A person who has received treatment for active TB or LTBI A person who has received an anti-TNFalpha treatment A person who has had a TST Pregnant women A person who has been diagnosed with a NTM infection

NTM population:

Inclusion criteria A person who is positive for NTM of interest confirmed by culture and identification;

Non-inclusion criteria A person who has been on antibiotic treatment for NTM; A person with confirmed active TB; A person with HIV; A person with a history of active TB; A person who have received treatment for LTBI; A person who is at high risk for LTBI Pregnant women.

Precision Population

Inclusion criteria:

A person previously enrolled in the Active TB, High Risk or Low Risk studies, or a blood donor.

Non-inclusion criteria An adult who was not previously enrolled in the Active TB, High Risk or Low Risk studies except for blood donors

For blood donors only:

A person who can be classified as being at increased risk for M. tuberculosis infection (and therefore LTBI) and/or for progression to active TB

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll persons with low to high risk factors for acquiring TB infection, persons with active TB disease, and persons with other types of Mycobacterial infections
Sampling Method: Non-Probability Sample
Enrollment: 2401 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Positive, negative, indeterminate for tuberculosis | One-time measurement through study completion for each participant, an average of 5 months.
  The VIDAS or comparator assays will qualitatively determine the presence or absence of Mycobacterial TB infection in a participant's blood. This measurement is based on the level of interferon gamma released after stimulation of T cells in blood.
Sensitivity and positive and negative percent agreement for the VIDAS TB IGRA assay with comparator assay | One-time measurement through study completion for each participant, an average of 5 months.
  Results obtained using the VIDAS assay will be compared with the results obtained from other methods.
Degree of Interference by nontuberculous mycobacteria for the VIDAS TB IGRA assay | One-time measurement through study completion for each participant, an average of 5 months.
  Persons with NTM will be tested using the VIDAS TB IGRA.
Measurement Precision of the VIDAS TB IGRA assay results | Triplicate measurement per sample through study completion, an average of 5 months.
  6- 4mL blood samples will be collected from each participant and tested using different VIDAS instruments.

CONTACTS AND LOCATIONS:
Overall Officials: David Pride, Principal Investigator — UC San Diego; Maria Gennaro, Principal Investigator — Rutgers University; Michael Lauzardo, Principal Investigator — University of Florida; Niaz Banaei, Principal Investigator — Stanford University; Nahed Ismail, Principal Investigator — University of Illinois Chicago; Daniel Hoft, Principal Investigator — St. Louis University; Charles Daley, Principal Investigator — National Jewish Health; Amanda Lopes, Principal Investigator — Lariboisière Hospital; Frederic Méchaï, Principal Investigator — Avicenne Hospital; Florence Doucet-Populaire, Principal Investigator — Antoine-Béclère Hospital; Elisabeth Botelho-Nevers, Principal Investigator — North Hospital
Locations (24):
- United States (7):
  - Stanford University, Palo Alto, California
  - UC San Diego, San Diego, California
  - Naional Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Illinois- Chicago, Chicago, Illinois
  - Saint Louis University, St Louis, Missouri
  - Rutgers University, Newark, New Jersey
- Brazil (2):
  - Universidade Federal de Mato Grosso do Sul (UFMS), Campo Grande
  - Universidade Federal Da Grande Dourados (UFGD), Dourados
- France (6):
  - Anti-TB center of Chambéry, Chambéry
  - Lapeyronie Hospital, Montpellier
  - Anti-TB center of Nanterre, Nanterre
  - Avicenne Hospital, Paris
  - Lariboisière Hospital, Paris
  - North Hospital, Saint-Etienne
- National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia
- Hinduja Hospital, Mumbai, India
- INMI L. Spallanzani, Rome, Italy
- Autonomous University of Baja California, Mexicali, Mexico
- South Africa (2):
  - TASK Applied Science, Delft Day Hospital Premises, Cape Town
  - University of Cape Town Centre for Lung Infection and Immunity, South Africa
- United Kingdom (3):
  - Evelina London Children's Hospital, London
  - Royal Free Hospital, London
  - St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No